CLINICAL TRIAL: NCT02433665
Title: Clinical Trial of a Novel Evidence-Based Formula for Customizing the Contrast Media Dose and Rate Administered During Multidetector-Row CT (MDCT) Scanning of the Abdomen and Pelvis
Brief Title: Customized Contrast Media Dose Clinical Trial
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow enrollment.
Sponsor: Duke University (Other)
Collaborators: Nemoto Kyorindo Co, Ltd. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: Pro00059984
Record Dates: First submitted 2015-04-24; First posted 2015-05-05 (Estimated); Results first posted 2020-06-16 (Actual); Last update posted 2020-06-16 (Actual); Status verified 2020-05

CONDITIONS: CT of the Abdomen and Pelvis With Contrast Material
MeSH Terms: interventions — Iopamidol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Fixed dose (Active Comparator): 100 of the first 200 subjects will be randomized to a fixed dose of contrast material.
  Interventions: Drug: Iopamidol
- Customized dose (Active Comparator): 100 of the first 200 subjects will be randomized to a customized dose of contrast material based on the experimental algorithm. The second group of 300 subjects will receive a customized dose of contrast material based on the experimental algorithm.
  Interventions: Drug: Iopamidol; Device: Mydose

INTERVENTIONS:
Drug: Iopamidol — Iopamidol is the contrast material being used for this study. 100 subjects will receive a fixed dose and rate (150 mL of iopamidol with a concentration of 300 mg of iodine/mL at an injection rate of 3 mL/sec for a total dose of 45 grams of iodine) and 400 subjects will be administered a customized dose and rate (X mL of iopamidol with a concentration of 300 mg of iodine/mL at an injection rate of X mL/sec for a total dose of X grams of iodine).
Device: Mydose — 400 subjects will receive a customized dose of contrast material (iopamidol) based on the experimental algorithm Mydose using a combination of subject parameters.
  Arms: Customized dose

SUMMARY:
1. To determine if a formula derived from PCA using specific patient parameters can be used to determine the individual contrast material dose and provide a more consistent level of vascular and parenchymal enhancement during MDCT scanning of the abdomen and pelvis.
2. Up to 500 adult patients referred for a "CT of the abdomen and pelvis with contrast material" will be recruited to participate in this trial. Single CT axial slices (n=2) will be obtained at the level of the L4 pedicle and the supra-acetabular pelvis using a field-of-view that includes all of the patient. From patient measurements (height, weight, body dimensions), a customized dose of contrast material will be specified according to the derived formula for 400 subjects. One hundred subjects will receive the usual fixed contrast dose.
3. Enhancement data in HU will be measured from the CT scans using manually-placed ROIs on the upper abdominal aorta, main portal vein and liver parenchyma, avoiding visible liver tumors, major blood vessels and artifacts, if present. This enhancement data will be used to determine the patient-to-patient variability.

DETAILED DESCRIPTION:
The next step is a single center, prospective clinical trial intended to test the hypothesis that a formula derived from PCA using specific subject parameters can be used to determine the individual contrast material dose and provide a more consistent level of vascular and parenchymal enhancement during MDCT scanning of the abdomen and pelvis.

500 subjects referred for a "CT of the abdomen and pelvis with contrast material" will be recruited to participate in this trial. Subjects in the first group of 200 will be randomized to either a fixed dose of contrast material (100 subjects) or a customized dose of contrast material based on the experimental algorithm (100 subjects). The second group of 300 subjects will receive a customized dose of contrast material based on the experimental algorithm. All of the subjects will be studied on a single CT scanner located in the Duke Cancer Center. After obtaining informed consent, the subjects will first undergo measurement of their height and weight on a dedicated pair of scales located in close proximity to the scanner.

The subjects will then be placed on the CT scan table in the supine position followed by the acquisition of scout digital radiographs in both the AP and ML projections. These digital scout radiographs are acquired routinely and used by the technologist to plan the scan. From these scout radiographs, single CT slices in the axial plane (n=2) will subsequently be obtained, one through the level of the L4 pedicle and the other through the supra-acetabular pelvis using a field-of-view that includes all of the subject. These slices are not part of the routine protocol but will be acquired using low radiation dose parameters. From these measurements (height, weight and specific body dimensions), a customized dose of contrast material will be specified according to the derived formula. Since the dose will be different in every subject, the rate will need to be adjusted as well. This will be accomplished by adjusting the rate so that the injection duration is the same in every subject. For example, if the specified contrast material dose is 100 mL and the injection duration is 25 seconds, the injection rate will be 4 mL/sec. If the specified contrast material dose is 125 mL and the injection duration is also 25 seconds, the injection rate will be increased to 5 mL/sec. Note that 100 subjects will receive a fixed dose and rate (150 mL of iopamidol with a concentration of 300 mg of iodine/mL at an injection rate of 3 mL/sec for a total dose of 45 grams of iodine) and 400 subjects will be administered a customized dose and rate (X mL of iopamidol with a concentration of 300 mg of iodine/mL at an injection rate of X mL/sec for a total dose of X grams of iodine) and. Also note that for the customized dose group, the maximum and minimum doses of contrast material will be 200 (75 gm iodine) and 75 (22.5 gm iodine) mL, respectively and the maximum and minimum injection rates will be 6 and 2 mL/sec, respectively. Because the injection rate in the customized group is variable, the nurse or technologist establishing intravenous access may choose to use a larger or small caliber angiocatheter than in the fixed group in order to accommodate a higher or lower injection rate, respectively. The caliber of the angiocatheter as well as the venous access site will be recorded along with the dose and rate of contrast material. The rate of administration of contrast material is controlled by a mechanical power injector furnished by Nemoto Kyorindo Co, Ltd. free of charge for use in this study.

ELIGIBILITY:
Inclusion Criteria:

* Patients referred for a CT of the Abdomen & Pelvis with Contrast Material

Exclusion Criteria:

* Younger than 18
* Pregnant
* Contraindication of iodinated contrast material
* Contraindication to a bolus injection
* Indication for biphasic exam (arterial + venous phases)
* Diffuse hepatic disease
* Subjects weighing more than 300 pounds

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 166 (Actual)
Dates: Start 2015-08; Primary Completion 2016-10-06 (Actual); Study Completion 2016-10-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniele Marin, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 10 enrolled subjects either screen failed or were withdrawn by the PI prior to randomization. Four subjects screen failed due to changes in their clinical orders prior to imaging. Six subjects were withdrawn by the PI due to patient scheduling conflicts.
Period: Overall Study
Arm/Group | Fixed Dose | Customized Dose
Started | 77 | 79
Completed | 77 | 79
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fixed Dose | Customized Dose | Total
Number analyzed (Participants) | 77 | 79 | 156
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.2 (13.6) | 61.7 (12) | 62.4 (12.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 30 | 62
  Male | 45 | 49 | 94
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 75 | 79 | 154
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 10 | 13 | 23
  White | 65 | 65 | 130
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Variability in Enhancement Data, Measured in Hounsfield Units (HU)
Time Frame: During CT scan, approximately 5 minutes
Measure: Mean (Standard Deviation); unit: Hounsfield Units (HU)
Arm/Group | Fixed Dose | Customized Dose
Number analyzed (Participants) | 77 | 79
Hounsfield Units (HU) | 199 (45) | 205 (50)
Statistical Analysis 1: Comparison: Fixed Dose vs Customized Dose; Test type: Non-Inferiority — The primary end point for this study was a comparison between fixed-dose and customized-dose contrast material injection CT protocols for vascular and parenchymal enhancement by using a noninferiority approach. The limit of noninferiority was set at 0.1 before the initiation of the study on the basis of a similar study that examined contrast media dose optimization for CT angiography examinations; p > 0.05, Mixed Models Analysis; Odds Ratio, log = 0.75, Standard Deviation 0.35

ADVERSE EVENTS:
Time Frame: 30 days from date of enrollment
Arm/Group | Fixed Dose | Customized Dose
All-Cause Mortality (participants affected / at risk) | 0/77 | 0/79
Serious Adverse Events (participants affected / at risk) | 0/77 | 0/79
Other Adverse Events (participants affected / at risk) | 0/77 | 0/79

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No